CLINICAL TRIAL: NCT00002104
Title: Placebo-Controlled Trial of Safety and Efficacy of Thalidomide in Patients With Infections Due to Mycobacterium and/or HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aaron Diamond AIDS Research Center (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 133A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-07

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections; Tuberculosis, Mycobacterium Infection
Keywords: Mycobacterium tuberculosis; Mycobacterium Infections; AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Mycobacterium Infections, Atypical; Thalidomide
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Tuberculosis; Mycobacterium Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Mycobacterium Infections, Nontuberculous | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
To demonstrate, in patients with tubercular or nontubercular mycobacterium infections with or without HIV infection, the safety of thalidomide use as judged by symptoms, physical exam, and studies of microbiologic, immunologic, hematologic, renal, and hepatic status. To demonstrate efficacy of the drug as judged by status of fever, nutrition, tuberculosis lesions, and immune responses.

DETAILED DESCRIPTION:
Patients are randomized to receive thalidomide or placebo orally at 9 PM the night before beginning anti-tuberculosis chemotherapy and continuing nightly for 7 nights. Patients are followed for 28 days. Patients are stratified according to HIV status and stage of HIV infection.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Positive AFB smear and/or culture for Mycobacterium tuberculosis, M. avium, or other mycobacterial infection, with or without documented HIV infection. NOTE:
* HIV-positive patients must have CD4 count < 500 cells/mm3 and be on antiretroviral therapy.
* One of the following manifestations:
* Temperature over 38 C on at least two occasions in the week prior to study entry.
* Recent weight loss of more than 5 kilograms.
* Pulmonary involvement of one or more lobes or involvement of other tissues due to tuberculosis or other mycobacterial infections, or symptomatic infections related to HIV status.
* Night sweats on two or more occasions in the week prior to study entry.

NOTE:

* Patients must be hospitalized men aged 18-65 and postmenopausal women to age 65. Anticipated requirement for hospitalization must be at least 10 days.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Neuropathy or other disorders with risk of neuropathy.

Required for HIV-positive patients if CD4 count < 500 cells/mm3:

* Antiretroviral therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Bellevue Hosp Ctr, New York, New York
  - Aaron Diamond AIDS Rsch Ctr / Rockefeller Univ, New York, New York